CLINICAL TRIAL: NCT02652182
Title: Short-term Air Pollution Exposure and In-hospital Outcomes in Patients With Acute Myocardial Infraction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nanjing Medical University (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jin Geng, MD, Nanjing Medical University
Other Study IDs: 20160006
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Air Pollution; Acute Myocardial Infarction; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with acute ST (S- and T-wave)-segment elevation myocardial infarction who received emergent percutaneous coronary intervention in Huai'an first people's hospital
- 2: patients with acute ST(S- and T-wave)-segment elevation myocardial infarction who received emergent percutaneous coronary intervention in Nanjing Drum Tower hospital

SUMMARY:
The aim of this study is to investigate whether or not short-term expose to air pollution is associated with in-hospital outcomes, such as mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Less than 12 hours after the onset of myocardial infarction symptoms
* Documented acute ST (S- and T-wave)-segment elevation myocardial infarction
* Received emergent percutaneous coronary intervention

Exclusion Criteria:

* Age under 18-year old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute ST (S- and T-wave)-segment elevation myocardial infarction who received emergent percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | in the phase of hospital stay, up to 30 days

SECONDARY OUTCOMES:
Length of hospital stay | in the phase of hospital stay, up to 30 days
ST (S- and T-wave) segment decreasing | within an hour after primary percutaneous coronary intervention
left ventricular function | in the phase of hospital stay, up to 30 days
  left ventricular ejection fraction in % and left ventricular end-diastolic diameter in mm, both are evaluated by echocardiography to assess the left ventricular function

CONTACTS AND LOCATIONS:
Locations (1):
- Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No